CLINICAL TRIAL: NCT05175560
Title: Baby Breathing Monitoring @Home
Status: Completed | Type: Observational
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Other Study IDs: ICBE-S-000608; NL79600.100.21 (Other: MEC-U)
Record Dates: First submitted 2021-12-06; First posted 2022-01-04 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Healty Babies; 3 Weeks - 3 Months Old
Keywords: Infants; physiology; behavior; respiration; sleep; unobtrusive monitoring; home setting
MeSH Terms: conditions — Behavior; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To give reassurance to parents, Philips would like to add algorithms to the NightOwl baby monitor to be able to measure baby behavior and physiology.

In this study, the investigators aim to investigate the applicability of in-house breathing algorithms, and to develop algorithms, for babies sleeping in a home setting.

The data collection will be divided in several sub-studies, either e.g. matching different development steps in the development of the algorithm or focusing on a specific baby population (e.g. specific age range). In general, babies will be monitored (audio, video, activity) for 24 -48 hours under their habitual sleeping conditions.

Step 1: 3 full data sets will be recorded of babies in bed aged 3 weeks to about 3-4 months, who are not able to turn over yet. Data will be analyzed and study set-up will be checked. Parents will be asked to keep a baby sleep diary and a questionnaire will be filled in at the start, with questions regarding the sleep behavior of their child. At the end, parents will be asked to fill in a questionnaire with sleep-related and feedback questions.

In step 2, 5 full data sets will be collected following the same procedure as step 1.

In step 3 12 full data sets will be collected following the same procedure as step 1.

After each step, the study setup including the algorithms, will be reviewed based on the obtained data. All modifications to this protocol will be submitted as amendments.

After step 1 and 2, the Mother and Child Care Business unit of Philips and other relevant stakeholders will be updated on the progress and findings by means of a (short) meeting and PowerPoint slides.

After step 3, a report will be written. The PowerPoint slides shared after Step 1 and 2 will be incorporated in this report.

DETAILED DESCRIPTION:
Procedures Phone call

During the Phone call the investigators will:

* explain the study setup
* explain the exclusion and inclusion criteria. The criteria will not be verified until visit 1.
* if the parents or caregivers agree, an appointment will be made for visit 1

  1. Home visit 1 - about 45 min

     During the first home visit the investigators will:

  <!-- -->

  1. a. make introductions;

  <!-- -->

  1. b. explain the study again, if necessary, and answer questions;

  1c. together with the subject's parents or caregivers sign the informed consent form belonging to this study;
* confirm the inclusion and exclusion criteria
* Complete the BISK questionnaire (investigator will ask questions to parent and report answers in CRF) 1d. Provide parents a baby sleep diary and instruct them to complete it; 1e. place the study setup in the room the baby mainly sleeps in; 1f. plan the second home visit. 2. During the study (2 consecutive days, including the nights) The setup will monitor the baby's bed, and the baby when the baby is in bed. After the setup is turned on, during Home Visit 1, it will record continuously for about two days (during day and night), until the investigator comes back to pick the setup up (see also Home Visit 2, below). The recording happens automatically; subject's parents or caregivers do not need to do anything with the setup.

The investigators will ask the parents or caregivers to keep a diary of the baby's (sleeping) behavior and to note information of behavior influencing the baby's sleep (e.g. baby being ill, not feeding well) during the recording period or if there was anything out of the ordinary with the setup (siblings fidgeting with it, power outings etc.).

In case of emergency, the recording can be stopped by pulling the electrical cord from the socket.

3. Home visit 2 - ~30 min

During the second home visit, the investigators will:

3a. ask how the study went, and if the parents or caregivers have any feedback for the investigators (close out questionnaire, investigator will ask questions to parent and report answers in CRF); 3b. review the sleep diary for omissions 3c. Check the end time and study setup 3d. pick up the test setup.

After completion of the participation, the investigator will notify the recruitment agency to arrange the compensation.

Devices used:

Survey/questionnaire: Baby diary and sleep related questions CE-approved non-medical device within intended use: Camera Non-medical device prototype: Bender, modified NightOwl video camera Other: PCs, Pole ( Monitor stand Generic, brand: König & Meyer 26785-018-56, commercially available)

ELIGIBILITY:
Inclusion Criteria:

Parents or caregivers :

* Have a baby aged >3 weeks to ~3-4 months (who is not yet able to role over; see exclusion criteria);
* Have a baby who sleeps in its own bed (i.e. different sleeping surface than parents; same room is allowed);
* Live in the Netherlands;.
* Are able to speak and read Dutch or English.

Exclusion Criteria:

Parents or caregivers

* with a baby who can already roll over (belly to back and back to belly);
* with a baby who is under supervision of an HCP because of health, feeding or developmental problems ;
* are unwilling or unable to provide informed consent on behalf of themselves, their baby and siblings;
* are unwilling or unable to comply with the study requirements;
* do not give permission to use their, or that of potential siblings, audio-video image data recorded during the study as described in the information letter and privacy notice;
* are not able to fill in the questionnaires and baby sleep diary.

Ages: 3 Weeks to 4 Months | Sex: All
Age Groups: Child
Study Population: healthy infants and their parents
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Can we measure baby behavior and physiology by camera and / or wearable? | through study completion, up to 1 year

SECONDARY OUTCOMES:
Can we measure breathing at all by camera when the baby is in bed? | up to 3 months
Can we measure when the baby is in and out of bed? | up to 3 months
Can we derive sleep stages from the data? | up to 3 months
Can we detect and / or interpret baby crying? | up to 3 months
Can we distinguish the baby (audio & movement) from other people near the bed (i.e. parents and/or siblings)? | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Renee Otte, dr, Principal Investigator — Philips Electronics Nederland B.V. acting through Philips CTO organization
Locations (1):
- Philips Research, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Coded data will be shared with Philips Mother and Child Care Business Unit : Questionnaires/diary, Activity data, Audio data, Video Data
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: the data will be shared after the data have been annotated and annotated data has been removed. Data will be available for maximum 20 years.

REFERENCES:
- [Background] Yue Sun, Wenjing Wang, Xi Long, Mohammed Meftah, Tao Tan, Caifeng Shan, Ronald M. Aarts, Peter H.N. de Widt; Respiration Monitoring for Premature Neonates in NICU; Appl. Sci. 2019, 9(23), 5246; https://doi.org/10.3390/app9235246
- [Background] Lorato I, Stuijk S, Meftah M, Kommers D, Andriessen P, van Pul C, de Haan G. Towards Continuous Camera-Based Respiration Monitoring in Infants. Sensors (Basel). 2021 Mar 24;21(7):2268. doi: 10.3390/s21072268. PMID 33804913
- [Background] Khan AU, Mikut R, Reischl M. A Benchmark Data Set to Evaluate the Illumination Robustness of Image Processing Algorithms for Object Segmentation and Classification. PLoS One. 2015 Jul 20;10(7):e0131098. doi: 10.1371/journal.pone.0131098. eCollection 2015. PMID 26191792
- [Background] Sadeh A. A brief screening questionnaire for infant sleep problems: validation and findings for an Internet sample. Pediatrics. 2004 Jun;113(6):e570-7. doi: 10.1542/peds.113.6.e570. PMID 15173539